CLINICAL TRIAL: NCT07035106
Title: I-WEAR: From ICU to Recovery - Evaluating the Feasibility and Usability of Bi-Weekly Health Summaries Using Wearables in Patients After Intensive Care Unit Treatment - A Pilot Study
Brief Title: I-WEAR: Evaluating Wearables and Health Summaries in ICU Survivors
Acronym: I-WEAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig Boltzmann Gesellschaft (Other)
Responsible Party: Principal Investigator, Akos Tiboldi, Principal Investigator, Ludwig Boltzmann Gesellschaft
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I-WEAR-PICS-1303-2025; DRP0200543 (Other Grant/Funding Number: European Union / Interreg Danube Region Programme)
Record Dates: First submitted 2025-05-24; First posted 2025-06-24 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Post-Intensive Care Syndrome (PICS); Critical Illness Recovery; Coronary Artery Disease
Keywords: Wearables; Health-related quality of life; ICU survivors; Digital health; Remote patient monitoring; System Usability Scale; SF-36; Bi-weekly health summary; Pilot study; PICS; Cardiovascular disease; Diabetes
MeSH Terms: conditions — postintensive care syndrome; Coronary Artery Disease; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1:1 into standard care, wearable use only, or wearable use with digital health summaries and optional counseling. There is no crossover between groups.
Masking Description: All participants and staff are aware of the assigned intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard care (No Intervention): Participants receive standard ICU follow-up care at the Medical University of Vienna without wearable devices or digital health tools.
- Wearables Only (Experimental): Participants receive wearable health monitoring devices (Garmin Vivosmart 5, Garmin Index S2 Smart Scale, Garmin Index BPM blood pressure monitor) and use the Fitrockr application to visualize and track their data. No counseling or bi-weekly summaries are provided.
  Interventions: Device: Wearable Health Monitoring
- Wearables + Summary + Counseling (Experimental): Participants receive the same wearable devices and Fitrockr app as the Wearables Only group. In addition, they receive bi-weekly automatically generated health summaries via email and have the option to book lifestyle consultations with a member of the study team via Webex.
  Interventions: Device: Wearable Health Monitoring; Behavioral: Digital Health Summary and Lifestyle Counseling

INTERVENTIONS:
Device: Wearable Health Monitoring — Participants receive a Garmin Vivosmart 5, Garmin Index S2 Smart Scale, and Garmin Index BPM blood pressure monitor for daily health tracking. Devices sync to the Fitrockr mobile application.
  Arms: Wearables + Summary + Counseling; Wearables Only
Behavioral: Digital Health Summary and Lifestyle Counseling — Participants receive bi-weekly health summaries via email generated from wearable data and may opt in to monthly video-based lifestyle consultations with trained study staff.
  Arms: Wearables + Summary + Counseling

SUMMARY:
This pilot study investigates the use of wearable health technology and bi-weekly digital health summaries in patients recovering from intensive care. Many patients experience physical, psychological, and cognitive challenges after an ICU stay, a condition known as Post-Intensive Care Syndrome (PICS). The study aims to evaluate the feasibility and usability of wearable devices-such as smartwatches, blood pressure monitors, and smart scales-for tracking recovery in real-world settings.

Participants will be randomly assigned to one of three groups: standard ICU follow-up care, wearable use only, or wearable use combined with bi-weekly health reports and optional lifestyle consultations. The study will assess participants' quality of life, experience using the technology, and adherence over a 6-month period. Results will inform the future use of digital tools in post-ICU care.

DETAILED DESCRIPTION:
I-WEAR is a single-center, non-invasive, randomized feasibility study conducted at the Medical University of Vienna in collaboration with the Ludwig Boltzmann Institute for Digital Health and Patient Safety. The study targets ICU survivors aged 18-65 years with prior ICU stays of ≥48 hours and comorbid diabetes mellitus and/or cardiovascular disease. The goal is to evaluate the feasibility and usability of wearable technologies and digital health reporting to enhance longitudinal care after ICU discharge.

Participants (n=60) are randomized into three groups:

Control group: Standard ICU follow-up care Intervention group 1: Wearables and app (smartwatch, scale, blood pressure monitor) Intervention group 2: Same wearables plus automated bi-weekly health summaries and optional health consultations via Webex Wearable devices include the Garmin Vivosmart 5 (tracking HRV, sleep, stress, and activity), the Garmin Index S2 Smart Scale, and the Garmin Index BPM blood pressure monitor. Data is aggregated via the Fitrockr application and stored in an ISO/IEC 27001-certified cloud environment in compliance with the EU General Data Protection Regulation (GDPR). Participants retain full control over data sharing, and pseudonymized data will be used for research purposes only.

The primary outcomes are feasibility (recruitment, retention, device adherence), and usability (System Usability Scale, qualitative interviews). Secondary outcomes include health-related quality of life measured via SF-36 at enrollment, mid-study (month 3), and study completion (month 6). Descriptive statistics and visualizations will summarize adherence and change trajectories. The study follows CONSORT 2010 guidelines for feasibility studies and includes a decision framework to inform whether to proceed with a definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years at the time of ICU admission
* ICU stay of at least 48 hours
* ICU discharge within the last 2 years
* Comorbidity of diabetes mellitus and/or chronic heart failure/coronary artery disease
* Written informed consent
* Access to a home internet connection and smartphone with internet and Bluetooth

Exclusion Criteria:

* Presence of a legal guardian
* No smartphone or internet access
* No cardiovascular disease/event and/or diabetes
* Implanted pacemaker or defibrillator
* Allergies to materials in the wearable devices
* Transfer from an ICU outside the Medical University of Vienna
* Homelessness
* Residence outside of Austria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Usability of Wearables in ICU Survivors | At 6 months after study enrollment
  Feasibility will be assessed by recruitment rate, retention rate, and adherence to wearable device use. Usability will be assessed using the System Usability Scale (SUS) at the end of the study.

SECONDARY OUTCOMES:
Change in Health-Related Quality of Life (HRQoL) | From enrollment (month 0) to study end (month 6)
  Measured using the SF-36 Version 2 questionnaire at baseline, mid-point (3 months), and end of study (6 months). Group-level and within-subject changes will be analyzed.
Acceptability of Lifestyle Counseling | Over 6-month intervention period
  Number and proportion of participants in intervention group 2 who schedule and attend at least one lifestyle counseling session.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Willschke, Ao. Univ. Prof. Dr., Study Director — Medical University of Vienna / Ludwig Boltzmann Institute for Digital Health and Patient Safety
Locations (1):
- Ludwig Boltzmann Institute Digital Health and Patient Safety, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to data protection regulations under the EU General Data Protection Regulation (GDPR). All data is pseudonymized and stored securely for internal analysis only. Future use of anonymized data for secondary research will require separate ethical approval and is not planned at this time.

REFERENCES:
- [Background] Pearson N, Naylor PJ, Ashe MC, Fernandez M, Yoong SL, Wolfenden L. Guidance for conducting feasibility and pilot studies for implementation trials. Pilot Feasibility Stud. 2020 Oct 31;6(1):167. doi: 10.1186/s40814-020-00634-w. PMID 33292770
- [Background] Teresi JA, Yu X, Stewart AL, Hays RD. Guidelines for Designing and Evaluating Feasibility Pilot Studies. Med Care. 2022 Jan 1;60(1):95-103. doi: 10.1097/MLR.0000000000001664. PMID 34812790
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Tison GH, Sanchez JM, Ballinger B, Singh A, Olgin JE, Pletcher MJ, Vittinghoff E, Lee ES, Fan SM, Gladstone RA, Mikell C, Sohoni N, Hsieh J, Marcus GM. Passive Detection of Atrial Fibrillation Using a Commercially Available Smartwatch. JAMA Cardiol. 2018 May 1;3(5):409-416. doi: 10.1001/jamacardio.2018.0136. PMID 29562087
- [Background] Bayoumy K, Gaber M, Elshafeey A, Mhaimeed O, Dineen EH, Marvel FA, Martin SS, Muse ED, Turakhia MP, Tarakji KG, Elshazly MB. Smart wearable devices in cardiovascular care: where we are and how to move forward. Nat Rev Cardiol. 2021 Aug;18(8):581-599. doi: 10.1038/s41569-021-00522-7. Epub 2021 Mar 4. PMID 33664502
- [Background] Duggan MC, Wang L, Wilson JE, Dittus RS, Ely EW, Jackson JC. The relationship between executive dysfunction, depression, and mental health-related quality of life in survivors of critical illness: Results from the BRAIN-ICU investigation. J Crit Care. 2017 Feb;37:72-79. doi: 10.1016/j.jcrc.2016.08.023. Epub 2016 Aug 31. PMID 27652496
- [Background] Desai SV, Law TJ, Needham DM. Long-term complications of critical care. Crit Care Med. 2011 Feb;39(2):371-9. doi: 10.1097/CCM.0b013e3181fd66e5. PMID 20959786
- [Background] Jackson JC, Pandharipande PP, Girard TD, Brummel NE, Thompson JL, Hughes CG, Pun BT, Vasilevskis EE, Morandi A, Shintani AK, Hopkins RO, Bernard GR, Dittus RS, Ely EW; Bringing to light the Risk Factors And Incidence of Neuropsychological dysfunction in ICU survivors (BRAIN-ICU) study investigators. Depression, post-traumatic stress disorder, and functional disability in survivors of critical illness in the BRAIN-ICU study: a longitudinal cohort study. Lancet Respir Med. 2014 May;2(5):369-79. doi: 10.1016/S2213-2600(14)70051-7. Epub 2014 Apr 7. PMID 24815803
- [Background] Ohtake PJ, Lee AC, Scott JC, Hinman RS, Ali NA, Hinkson CR, Needham DM, Shutter L, Smith-Gabai H, Spires MC, Thiele A, Wiencek C, Smith JM. Physical Impairments Associated With Post-Intensive Care Syndrome: Systematic Review Based on the World Health Organization's International Classification of Functioning, Disability and Health Framework. Phys Ther. 2018 Aug 1;98(8):631-645. doi: 10.1093/ptj/pzy059. PMID 29961847
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] Mikkelsen ME, Still M, Anderson BJ, Bienvenu OJ, Brodsky MB, Brummel N, Butcher B, Clay AS, Felt H, Ferrante LE, Haines KJ, Harhay MO, Hope AA, Hopkins RO, Hosey M, Hough CTL, Jackson JC, Johnson A, Khan B, Lone NI, MacTavish P, McPeake J, Montgomery-Yates A, Needham DM, Netzer G, Schorr C, Skidmore B, Stollings JL, Umberger R, Andrews A, Iwashyna TJ, Sevin CM. Society of Critical Care Medicine's International Consensus Conference on Prediction and Identification of Long-Term Impairments After Critical Illness. Crit Care Med. 2020 Nov;48(11):1670-1679. doi: 10.1097/CCM.0000000000004586. PMID 32947467
- See also: Official study project page of the DIGI4Care - Transforming patient journeys through digital innovation in healthcare across the Danube Region — https://interreg-danube.eu/projects/digi4care
- See also: Official study project page from the Ludwig Boltzmann Institute for Digital Health and Patient Safety — https://dhps.lbg.ac.at/forschung/digital-tools/digi4care/?lang=en